CLINICAL TRIAL: NCT02010021
Title: Presurgical Treatment With Letrozole in Patients With Early-stage Breast Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Gary Schwartz, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: D13236
Record Dates: First submitted 2013-11-22; First posted 2013-12-12 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; postmenopausal; letrozole; RAD001; Everolimus
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: 10 subjects received no presurgical therapy, and then 7 subjects received presurgical letrozole.
  This is a sequential model because the results from Arm A determined the sample size for Arm B. Tumors from each of the 10 untreated patients in Arm A showed induction of AKT activation with RAD001 treatment. Based on these results, we determined that a sample size of seven patients from Arm B would be adequate to detect a significant effect (p≤0.05) of presurgical Letrozole on RAD001-induced changes in phospho-AKT levels with 80% power (calculated using uncorrected chi-squared statistic).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No drug treatment (No Intervention): Post-menopausal women with stage I-III breast cancer will have surgical resection of tumor and tumor tissue will be used to study cell growth signaling pathways ex-vivo.
- Letrozole-presurgical (Active Comparator): Patients will receive Letrozole for 10-21 days prior to surgical resection of tumor tissue. This tissue will be used ex-vivo to study cell growth signaling pathway. The results will be compared to arm of the study with no intervention.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Patients will receive Letrozole for 10-21 days prior to surgical resection of tumor tissue. This tissue will be used ex-vivo to study cell growth signaling pathway. The results will be compared to arm of the study with no intervention.
  Other Names: Femara
  Arms: Letrozole-presurgical

SUMMARY:
Some tumors use estrogen in the body to assist with growth. Letrozole is a drug that is prevents cells from producing estrogens. This should assist with the slowing of growth of tumor cells. Letrozole also promotes cell destruction by inhibiting a cellular destruction pathway.

The objectives of this study will look at the differences between the cellular destruction pathway before and after letrozole use, and the differences in the cellular destruction pathway in participants that have received letrozole versus those who did not. The study will also look at a gene in all participants called Ki67. This gene is associated with the rate of tumor cell growth. The study will measure the levels of Ki67 and compare them to the amount of activation of the cellular destruction pathway.

Participants in this study will have undergone a diagnostic biopsy of their breast tissue.

In order to meet these objectives, one group of participants (Arm A) will not receive letrozole. Tissue leftover from their diagnostic biopsy will be treated with everolimus (RAD001) in the laboratory and the effects of this drug on the cellular destruction pathway will be studied.

The other group of participants (Arm B) will take letrozole for a minimum of 10 and maximum of 21 days. They will have a second tumor sample taken as part of their surgical procedure completed to remove the tumor tissue. Any differences in the cellular destruction pathway before and after exposure to letrozole will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Histologic Documentation of invasive breast cancer by core needle or incisional biopsy. Excess baseline biopsy tumor tissue sufficient to make three 5-micron sections must be available for molecular analyses as part of this study.
* The invasive cancer must be estrogen receptor alpha (ER)-positive, with ER staining present in greater than 50% staining of invasive cancer cells by IHC.
* The invasive cancer must be human epidermal growth factor receptor 2 (HER2) negative (IHC 0-1+, or with a fluorescence in situ hybridization (FISH) ratio of <1.8 if IHC is 2+ or if IHC has not been done).
* Clinical stage I-III invasive breast cancer with the intent to treat with surgical resection of the primary tumor. Tumor must be ≥ 2cm to provide adequate tissue.
* Patients with multi-centric or bilateral disease are eligible if the target lesions meet the other eligibility criteria. Samples from all available tumors are requested for research purposes.
* Women ≥ age 18, for whom adjuvant treatment with an aromatase inhibitor would be clinically indicated. Women must be either post-menopausal, or pre-menopausal having undergone oophorectomy.
* Patients must meet the following clinical laboratory criteria:

Absolute neutrophil count (ANC)≥ 1000/mm3 and platelet count ≥ 75,000/mm3. Total bilirubin ≤ 1.5 X the upper limit of normal range (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.

- Ability to give informed consent.

Exclusion Criteria:

* Prior endocrine therapy for any histologically confirmed cancer is not allowed. Prior endocrine therapy that was administered ≥ 5 years ago for the prevention of breast cancer in patients with no history of breast cancer is allowed.
* Systemic drug treatment to induce ovarian suppression if woman is pre-menopausal.
* Any other neoadjuvant therapy for breast cancer (i.e., treatment with any other anti-cancer agent besides Letrozole (10-21)days before surgical resection of the primary tumor).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Schwartz, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Yang W, Schwartz GN, Marotti JD, Chen V, Traphagen NA, Gui J, Miller TW. Estrogen receptor alpha drives mTORC1 inhibitor-induced feedback activation of PI3K/AKT in ER+ breast cancer. Oncotarget. 2018 Jan 15;9(10):8810-8822. doi: 10.18632/oncotarget.24256. eCollection 2018 Feb 6. PMID 29507656

RESULTS

PARTICIPANT FLOW:
Groups:
- No Drug Treatment: Post-menopausal women with stage I-III breast cancer with surgical resection of tumor and tumor tissue will be used to study cell growth signaling pathways ex-vivo.
- Letrozole-presurgical: Patients received Letrozole for 10-21 days prior to surgical resection of tumor tissue. This tissue was used ex-vivo to study cell growth signaling pathway. The results will be compared to arm of the study with no intervention.
Period: Overall Study
Arm/Group | No Drug Treatment | Letrozole-presurgical
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Drug Treatment | Letrozole-presurgical | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Mean (Full Range); unit: years] | 65.6 [49 to 78] | 64.9 [55 to 77] | 65.3 [49 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, not Hispanic | 10 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Receptor Substrate 1 (IRS-1) / Phosphoinositide 3-kinase (PI3K) / Serine-threonine Protein Kinase (AKT) Pathway Activation
Description: The Primary Endpoint is to determine the effect of ex vivo mTORC1 inhibition with everolimus (RAD001) on IRS-1/PI3K/AKT pathway activation (as measured by phospho-AKT-T308 and phospho-AKT-S473) in ER+/human epidermal growth factor receptor 2 (HER2)- breast tumors treated with presurgical letrozole compared to ER+/HER2- breast tumors not treated with presurgical therapy.
Time Frame: baseline and surgery, approximately 30 days
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | No Drug Treatment | Letrozole-presurgical
Number analyzed (Participants) | 10 | 7
% change
  phospho-AKT-T308 | 388 (623) | -10 (38)
  phospho-AKT-S473 | 157 (35) | 135 (91)

2. Secondary Outcome: Percentage of Ki67 Score
Description: The Secondary Endpoint is to compare tumor cell proliferation as measured with the Ki-67 assay in breast cancer specimens taken before and at the time of surgery, comparing specimens of patients treated with presurgical letrozole and specimens of patients who did not receive presurgical letrozole. The secondary endpoint is Ki67 score, as determined by the percentage of Ki67+ tumor cells identified by immunohistochemistry.
  Whole slides were scanned at 40x (Aperio AT2, Leica Biosystems), and automated Ki67 analysis (percent positive nuclei) was determined using the Aperio ImageScope (v12.3.1.60002, Leica Biosystems) nuclear v9 algorithm. As recommended by the International Ki67 in Breast Cancer Working Group, 3 high-power microscopic fields were selected for analysis to represent the spectrum of staining present on the whole tissue section, and a minimum of 500 malignant invasive cells were score
Time Frame: baseline and surgery, approximately 30 days
Measure: Mean (Full Range); unit: change in % of Ki67+ tumor cells
Arm/Group | No Drug Treatment | Letrozole-presurgical
Number analyzed (Participants) | 10 | 7
change in % of Ki67+ tumor cells | -7.462 [-31.025 to 7.575] | -21.309 [-42.175 to -2.875]

ADVERSE EVENTS:
Time Frame: One month
Arm/Group | No Drug Treatment | Letrozole-presurgical
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT02010021/Prot_SAP_000.pdf